CLINICAL TRIAL: NCT03579810
Title: Impact of a Pedagogical Intervention on Children Cardiovascular Risk Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Cardioinfantil Instituto de Cardiología (Other)
Collaborators: Instituto Colombiano para el Desarrollo de la Ciencia y la Tecnología (COLCIENCIAS) (Other Government)
Responsible Party: Principal Investigator, CespedesJ_PI, Head of the Pediatric Service, Fundación Cardioinfantil Instituto de Cardiología
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IM-564-2012
Record Dates: First submitted 2018-06-26; First posted 2018-07-09 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Cardiovascular Health
Keywords: Behavioral Modification; Health Community; Community Intervention; Prevention; Education Intervention; Cardiovascular Health; Colombia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational (Experimental): An education intervention was implemented in 5 schools including 516 children, 360 parents and 240 teachers.
  The Pedagogical Intervention last two and a half years. In children, the intervention included class activities (1/week) and the use of educational materials for the development of pedagogical activities (posters and educative guide).
  In parents included 3 workshops/year (2 hours each) about the areas of the intervention; sending healthy notes (1/month) and celebration of healthy family day (1/year).
  In teachers included 3 workshops/year (2 hours each) about the areas of the intervention; planning and realization of pedagogical activities to develop with the students (1/week) and follow-up visits to school (1/month).
  Interventions: Other: Investigational
- Control (Active Comparator): The control group consisted of 4 schools including 354 children, 305 parents and 110 teachers.
  The activities in control group last two and a half years. Children received the standard curriculum in health and physical activity of the national Ministry of Education.
  In parents and teachers included 3 workshops/year (2 hours each) about the first aid and accident prevention.
  Interventions: Other: Control

INTERVENTIONS:
Other: Investigational — The educational intervention helped to increase the knowledge of attitudes, and habits of healthy lifestyle in children, parents and teachers and it was based on health promotion models and social cognitive theory, to be articulated with the Institutional Educational Project through the pedagogical component that integrates three areas, physical activity, healthy eating, and the knowledge of the body and the heart with the dynamics of the educative community.
  The program covered self-care of the body and heart, healthy diet, and physical activity
  Arms: Investigational
Other: Control — The control group did not receive an educational intervention in areas of physical activity, healthy eating, and the knowledge of the body and the heart. Instead, children received the standard curriculum in health and physical activity of the national Ministry of Education.
  Arms: Control

SUMMARY:
In Bogotá, Colombia, the Fundación Cadioinfantil performed a randomized and controlled community trial, to evaluate the impact of a pedagogical intervention (PI) on cardiovascular health towards an active lifestyle and healthy eating in 9 schools of the city, including children from kindergarten to second grade of elementary school, their parents and teachers.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is a leading cause of mortality worldwide and Colombia is not an exception. Epidemiological studies have demonstrated that CVD risk factors are identifiable in childhood and they are predictor of CDV risk in adulthood. Worldwide, CDV primary prevention that begins in childhood is identified as a strategy that decreases the burden of this disease.

Programs developed in educational communities (EC), that include in their planning and implementation students, teachers and parents, with training to food personnel, are the most effective strategies to create healthy school environments and reduce the burden of chronic diseases. However recent studies that evaluate physical activity through accelerometers have not shown effectiveness.

In 2009, the Si! program and Fundación CardioInfantil performed a randomized and controlled community trial in facilities of the Colombian Family welfare Institute, ICBF, from Usaquen locality in Bogotá, finding that a pedagogical intervention (PI) in preschool children, their parents and teachers is effective in improving knowledge, attitudes and habits towards an active lifestyle and healthy diet.

The construction of the proposed intervention is based on the best available evidence about programs, policies and practices that positively impact in healthy eating and physical activity habits in EC.

The objectives of this project are to evaluate changes in healthy foods consumption and energy expenditure in children from kindergarten to second grade of elementary school that receives pedagogical intervention (PI) adapted to its context, compared to another EC that develops its habitual curriculum. In addition, this study evaluates changes on cardiovascular risk factors in children. Also, it evaluates changes in healthy foods consumption in their parents and teachers.

ELIGIBILITY:
Inclusion Criteria:

* Private schools located in the urban area of Bogotá
* Schools with an appropriate physical activity space and infrastructure.
* Schools that allow the study conduction.

Exclusion Criteria:

* Schools that have received interventions of more than 1 month in healthy habits (nutrition and / or physical activity) during the year prior to the start of the study.
* Schools that plan to receive interventions of more than 1 month in healthy habits (nutrition and / or physical activity) during the time of follow-up of the study.
* Schools with a history of annual dropout of their students or teachers greater than 10%.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 870 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in active energy expenditure in children | Baseline and 2.5 years
  The energy expenditure (Kilocalories/day), in children from Kindergarten to grade 2 of elementary school, generated by physical activity was evaluated using accelerometers during 4 consecutive days, 24hours/day (2 weekend days and two schooldays) through an Actiheart® 4 type accelerometer.
  Possible differences between changes in active energy expenditure means was assessed using test t-test. Multi-variable models were performed to adjust for potential con-founders.
Changes in healthy foods consumption in children | Baseline and 2.5 years
  A food frequency survey (ENSIN 2010) was used in children from Kindergarten to grade 2 of elementary school.
  Healthy foods consumptions were defined as the accomplishment of 3-4 of the 4 measured components (intake of Fruits and vegetables ≥3 times a day, Fiber: ≥3 times a day, Fish: ≥2 times a week, Sugary beverages: ≤ 1 time a day).
  Possible differences between changes in the proportion of children with healthy foods consumption was assessed using chi2 test. Multi-variable models were performed to adjust for potential con-founders.

SECONDARY OUTCOMES:
Changes in the Body Mass Index in children | Baseline and 2.5 years
  Using the Quetelet index, that considers the BMI as the relationship between the body weight given in kg and the square size taken in meters.
  Possible differences between changes in BMI means was assessed using test t-test. Multi-variable models were performed to adjust for potential con-founders.
Changes in the perimeter of the waist in children | Baseline and 2.5 years
  Using a tape measure on the skin just above the iliac crest, in feet position. Possible differences between changes in perimeter of the waist means was assessed using test t-test. Multi-variable models were performed to adjust for potential con-founders.
Changes in total cholesterol in children | Baseline and 2.5 years
  Possible differences between changes in total cholesterol means was assessed using test t-test. Multi-variable models were performed to adjust for potential con-founders.
Changes in triglycerides in children | Baseline and 2.5 years
  Possible differences between changes triglycerides means was assessed using test t-test. Multi-variable models were performed to adjust for potential con-founders
Changes in fasting glycemia in children | Baseline and 2.5 years
  Possible differences between changes in fasting glycemia means was assessed using test t-test. Multi-variable models were performed to adjust for potential con-founders
Change in blood pressure in children | Baseline and 2.5 years
  Three measurements were made using a standardized technique. Possible differences between changes in both systolic and diastolic blood pressure means was assessed using test t-test. Multi-variable models were performed to adjust for potential con-founders.
Changes in the consumption of healthy foods in teachers | Baseline and 2.5 years
  A food frequency survey (ENSIN 2010) was used in teachers. Healthy foods consumptions were defined as the accomplishment of 3-4 of the 4 measured components (intake of Fruits and vegetables ≥3 times a day, Fiber: ≥3 times a day, Fish: ≥2 times a week, Sugary beverages: ≤ 1 time a day).
  Possible differences between changes in the proportion of teachers with healthy foods consumption was assessed using chi2 test. Multi-variable models were performed to adjust for potential con-founders.
Changes in the consumption of healthy foods in parents | Baseline and 2.5 years
  A food frequency survey (ENSIN 2010) was used in parents. Healthy foods consumptions were defined as the accomplishment of 3-4 of the 4 measured components (intake of Fruits and vegetables ≥3 times a day, Fiber: ≥3 times a day, Fish: ≥2 times a week, Sugary beverages: ≤ 1 time a day).
  Possible differences between changes in the proportion of parents with healthy foods consumption was assessed using chi2 test. Multi-variable models were performed to adjust for potential con-founders.

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Cespedes, MD, Principal Investigator — Fundación Cardioinfantil Instituto de Cardiología
Locations (1):
- Fundacion Cardioinfantil Instituto de Cardiologia, Bogotá, Bogota D.C., Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cespedes J, Briceno G, Farkouh ME, Vedanthan R, Baxter J, Leal M, Boffetta P, Woodward M, Hunn M, Dennis R, Fuster V. Targeting preschool children to promote cardiovascular health: cluster randomized trial. Am J Med. 2013 Jan;126(1):27-35.e3. doi: 10.1016/j.amjmed.2012.04.045. Epub 2012 Oct 9. PMID 23062403
- [Derived] Neil-Sztramko SE, Caldwell H, Dobbins M. School-based physical activity programs for promoting physical activity and fitness in children and adolescents aged 6 to 18. Cochrane Database Syst Rev. 2021 Sep 23;9(9):CD007651. doi: 10.1002/14651858.CD007651.pub3. PMID 34555181